CLINICAL TRIAL: NCT04103619
Title: Energy-Based Lower Eyelid Rejuvenation - Proof of Concept for InMode AccuTite With or Without Morpheus8
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InMode MD Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DO608677A
Record Dates: First submitted 2019-09-23; First posted 2019-09-25 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2022-01

CONDITIONS: Periorbital Edema
MeSH Terms: conditions — Orbital Cellulitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- AccuTite (Active Comparator): 15 patients will receive AccuTite treatment only
  Interventions: Device: AccuTite
- AccuTite & Morpheus 8 Arm (Active Comparator): 15 patients will receive AccuTite and Morpheus8 treatment and additional 2 monthly Morpheus8 treatments
  Interventions: Device: AccuTite + Morpheus 8

INTERVENTIONS:
Device: AccuTite — Subjects will undergo treatment with AccuTite
  Arms: AccuTite
Device: AccuTite + Morpheus 8 — Subjects will undergo treatment with AccuTite and Morpheus 8
  Arms: AccuTite & Morpheus 8 Arm

SUMMARY:
1. To establish clinical efficacy, safety and patient satisfaction of reducing lower eyelid convexities or "bags" and/or malar crescents (festoons) with catheter-based injectable RF (InMode AccuTite) and variable depth Fractional RF Microneedle skin rejuvenation (InMode Morpheus8).
2. To determine the relative effectiveness of dual-modality treatment (AccuTite + Morphues8 initial treatment followed by two consecutive Morpheus8 treatments 1 month apart) versus single modality treatment (AccuTite only)

DETAILED DESCRIPTION:
This prospective study is intended to evaluate the efficacy of radio frequency energy in reducing lower eyelid convexities or "bags" and/or malar crescents (festoons) with RFAL (InMode AccuTite) and variable depth Fractional RF resurfacing skin rejuvenation (InMode Morpheus8).

1. 15 patients will receive AccuTite treatment only (7-8 patients per arm at each of the two study sites)
2. 15 patients will receive AccuTite and Morpheus8 treatment and additional 2 monthly Morpheus8 treatments (7-8 patients per arm at each of the two study sites) Treatment areas include: periorbital zones with Morpheus8/Lower Eyelid with Accutite

ELIGIBILITY:
Inclusion Criteria:

* Adult females and males between the ages of 29-75 inclusive, having minimum level 1 for convexity for both lower eyelids.
* The patients should understand the information provided about the investigative nature of the treatment, possible benefits, and side effects, and sign the Informed Consent Form, (including the permission to use photography).
* The patients should be willing to comply with the study procedure and schedule, including the follow-up visit, and will refrain from using any other aesthetic treatment methods for the last 6 months and during the entire study period.

Exclusion Criteria:

* - Grade 3 lower eyelid convexity
* Grade 3 festoonage
* Prior lower eyelid fat removal (transconjunctival, transcutaneous)
* Prior lower eyelid skin resection
* Full-field or fractional laser skin resurfacing of lower eyelids in the past 24 months
* Tear trough, suborbital, midface filler injections in the past 24 months
* Neuromodulator treatment of crow's feet area in the past 12 months
* Lower eyelid malposition (rounding, retraction, ectropion, laxity)
* Meige syndrome
* Significant negative vector lower eyelid
* Pacemaker or internal defibrillator, or any other active electrical implant anywhere in the body.
* The Handpiece should be used at least 1cm away from cochlear implants in the ear.
* Superficial permanent implant in the treated area such as metal plates and screws, metal piercing, silicone implants or an injected chemical substance.
* Current or history of skin cancer (remission of 5 years), or current condition of any other type of cancer, or pre-malignant moles.
* Severe concurrent conditions, such as cardiac disorders, epilepsy, uncontrolled hypertension, and liver or kidney diseases.
* Pregnancy and nursing.
* History of bleeding coagulopathies or the use of anticoagulants.
* Impaired immune system due to immunosuppressive diseases such as AIDS and HIV or use of immunosuppressive medications.
* Poorly controlled endocrine disorders, such as diabetes or thyroid dysfunction and hormonal virilization.
* Any active condition in the treatment area, such as sores, psoriasis, eczema, and rash.
* History of skin disorders, keloids, abnormal wound healing, as well as very dry and fragile skin.
* Use of Isotretinoin (Accutane®) within 6 months prior to treatment.
* Any surgery or treatment such as laser or chemicals in the treated area within 3-6 months prior to treatment or before complete healing.
* Allergies, in particular to anesthesia.
* Mental disorders such as Body Dysmorphic Disorder (BDD).
* Monovision (single seeing eye)
* Corneal transplant
* Severe dry eyes
* As per the practitioner's discretion, refrain from treating any condition that might make it unsafe for the patient.

Ages: 29 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2021-12-13 (Actual)

PRIMARY OUTCOMES:
Correct identification at baseline and post treatment pictures | Change from baseline at 3 and 6 months
  Correct identification of the 3 and 6 Months post last treatment photographs from the baseline by at least two of the three blinded reviewers in 75% of the subjects.
Change in lower eyelid convexity scale | Change from baseline at 3 and 6 months
  Investigator assessment of the Lower eyelid convexity scale (based on right and left lateral photography assessments with Canfield Scientific imaging) at 3 and 6 months follow up visit and compared to the baseline, as follows: 0 = flat lower eyelid
  1. = mild convexity lower eyelid
  2. = moderate convexity lower eyelid
  3. = severe convexity lower eyelid
Change in Festoonage scale | Change from baseline at 3 and 6 months
  Investigator assessment of the Festoonage scale (based on photography assessments with Canfield Scientific imaging TBD) at 3 and 6 months follow up visit and compared to the baseline, as follows: 0 = no skin fold at or below inferior orbital rim
  1. = single skin fold at or below inferior orbital rim
  2. = double skin fold at or below inferior orbital rim
  3. = triple skin fold at or below inferior orbital rim
Subject assessment of satisfaction | Change from baseline at 3 and 6 months
  Subject assessment of satisfaction will be filled out by subjects using a 5-points
  Likert scale at 3 and 6 months follow up, as follows:
  +2 = Very satisfied; +1 = Satisfied; 0 = Indifferent; -1 = Disappointed; -2 = Very disappointed

CONTACTS AND LOCATIONS:
Overall Officials: David Holcomb, MD, Principal Investigator — Holcomb Kreithen Plastic Surgery and MedSpa; Richard Gentile, MD, Principal Investigator — Gentile Facial Plastic and Aesthetic Laser Center
Locations (2):
- United States (2):
  - David Holcomb, Sarasota, Florida
  - Gentile Facial Plastic and Aesthetic Laser Center, Youngstown, Ohio